CLINICAL TRIAL: NCT01551602
Title: Clinical Study of AK159 in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AK159 I-1
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2012-01

CONDITIONS: Osteoporosis
Keywords: AK159; teriparatide acetate
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (11):
- AK159 SD 1 (Experimental): Single administration of AK159 dose level 1
  Interventions: Drug: AK159
- AK159 SD 2 (Experimental): Single administration of AK159 dose level 2
  Interventions: Drug: AK159
- AK159 SD 3 (Experimental): Single administration of AK159 dose level 3
  Interventions: Drug: AK159
- AK159 SD 4 (Experimental): Single administration of AK159 dose level 4
  Interventions: Drug: AK159
- MN-10-T SD (Active Comparator): Single administration of MN-10-T
  Interventions: Drug: MN-10-T
- AK159 MD 1 (Experimental): Multiple administration of AK159 dose level 1
  Interventions: Drug: AK159
- AK159 MD 2 (Experimental): Multiple administration of AK159 dose level 2
  Interventions: Drug: AK159
- AK159 MD 3 (Experimental): Multiple administration of AK159 dose level 3
  Interventions: Drug: AK159
- AK159 MD 4 (Experimental): Multiple administration of AK159 dose level 4
  Interventions: Drug: AK159
- MN-10-T MD (Active Comparator): Multiple administration of MN-10-T
  Interventions: Drug: MN-10-T
- Placebo MD (Placebo Comparator): Multiple administration of placebo AK159
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK159 — transdermal administration of teriparatide acetate
  Arms: AK159 MD 1; AK159 MD 2; AK159 MD 3; AK159 MD 4; AK159 SD 1; AK159 SD 2; AK159 SD 3; AK159 SD 4
Drug: MN-10-T — subcutaneous administration of teriparatide acetate
  Arms: MN-10-T MD; MN-10-T SD
Drug: Placebo — Multiple administration of placebo AK159
  Arms: Placebo MD

SUMMARY:
The objective of this study is to investigate the pharmacokinetics, safety, and tolerability of AK159 administered to healthy postmenopausal women.

DETAILED DESCRIPTION:
This study consists of Part 1 and Part 2. <Part 1> Part 1 will be conducted according to a single-centre, randomized, single-dose, 3-period, 5-treatment alternating crossover design in two groups of healthy post-menopausal women The pharmacokinetics, safety, and tolerability of a single dose of AK159 (4 levels) will be investigated versus teriparatide acetate for injection as a control.

<Part 2> Part 2 will be conducted according to a multiple-centre, randomized, double-blind, placebo-controlled, repeated dose parallel design of healthy post-menopausal women The pharmacokinetics, safety, and tolerability of AK159 (4 levels) for 8 weeks will be investigated versus teriparatide acetate for injection and placebo as controls. Pharmacokinetics, safety, and tolerability following long-term application will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal ethnic Japanese women; At least 45 years of age at the time consent is obtained; and Give voluntary consent in writing with a sufficient understanding of the study.

Exclusion Criteria:

* Clinical abnormality identified in the laboratory tests
* Weight < 40.0 kg
* Body mass index < 17.5 or >=30.5
* History of disease of the kidneys, liver, heart, brain, or other organ that makes them ineligible as subjects
* Previously received radiation treatment potentially affecting bone
* Systolic blood pressure < 90 mmHg
* QTc exceeds 470 msec in a 12-lead electrocardiography
* Serum calcium level exceeding 10.4 mg/dL
* History of contact dermatitis or skin disease potentially compromising study evaluation
* Used drugs which impact bone metabolism in the 8-week period preceding investigational product administration
* Used a bisphosphonate;
* Used a teriparatide product;

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of teriparatide | up to 6 hours after single and repeated administration
Peak Plasma Concentration (Cmax) of teriparatide | up to 6 hours after single and repeated administration
Number of Participants with Adverse Events, Vital signs, ECG parameters, and 24-hour ECG holter recording (for Part 2 of the study). | up to 24 hours after single and repeated administration

SECONDARY OUTCOMES:
Change from Baseline in bone turnover markers within 24 hrs at each administration
Residual teriparatide in the patch after application

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Fukuoka
  - Kumamoto
  - Tokyo